CLINICAL TRIAL: NCT06525064
Title: Health-E You/Salud iTu: Pre-visit Mobile Health App for Male Adolescents to Promote Adolescent-centered Sexual & Reproductive Healthcare Receipt
Brief Title: Health-E You Efficacy Trial for Male Adolescents
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: IRB00424416; R01HD109141 (NIH)
Record Dates: First submitted 2024-07-18; First posted 2024-07-29 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Sexually Transmitted Diseases; Sexual Health; Reproductive Health
Keywords: male adolescent; condom use; mhealth
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Intervention Model Description: This study will use a cluster-randomized stepped-wedge design that is a type of one-way crossover design. Under this design, each clinic will start the study under the control condition that involves standard usual care, and end the study in the intervention condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): When clinics are in the control condition, patients will receive usual care. Before the visit eligible participants will receive a weblink to study information, and if agree to participate, the survey. The participants will not be presented Health-E You content and clinicians will not receive output to prime the visit; the participants will receive usual care as typical. Previously enrolled control males will not be enrolled during intervention periods to maintain the research study's integrity.
- Intervention Group (Experimental): When clinics are in the intervention condition, all patients presenting for any reason will get a study weblink 24 hours before the visit; walk-ins will get a study link code in clinic. If the participants agree to participate and meet study criteria, the participants will get a survey link and then Health-E You content to complete before the visit. Previously enrolled males will not be enrolled again to maintain the research study's integrity. Thus, participants will only have one opportunity for administration to the Health-E You app.
  Participants will be considered to have completed the Health-E You app if the participants answer all of the app's initial tailoring questions and receive recommendations for SRH topics to discuss with the clinician. As a technology-based intervention, no direct interactions with interventionists with participants are required.
  Interventions: Other: Health-E You app

INTERVENTIONS:
Other: Health-E You app — When clinics are in the intervention condition, all patients presenting for any reason will get a study weblink 24 hours before the visit; walk-ins will get a study link code in clinic. If the participants agree to participate and meet study criteria, the participants will get a survey link and then Health-E You content to complete before the visit. Previously enrolled males will not be enrolled again to maintain the research study's integrity. Thus, participants will only have one opportunity for administration to the Health-E You app.
  Participants will be considered to have completed the Health-E You app if the participants answer all of the app's initial tailoring questions and receive recommendations for SRH topics to discuss with the clinician. As a technology-based intervention, no direct interactions with interventionists with participants are required.
  Arms: Intervention Group

SUMMARY:
This study will involve evaluating Health-E You/Salud ìTu™, a web-based, pre-visit mobile app designed to support adolescent male youth and his clinicians in discussing sexual and reproductive health (SRH) topics and care. It will test its efficacy among male patients in clinical settings using a stepped wedge cluster randomized controlled trial design.

DETAILED DESCRIPTION:
Health-E You is a pre-visit, web-based mobile app designed to support an adolescent male youth and his clinician in discussing SRH topics and care. It is shared with an adolescent patient prior to a clinic visit, and contains initial questions that subsequently provide the patient with individually-tailored health information. In addition, the app provides relevant information to the clinician on patients' SRH to optimize the time together as part of the visit. In total, the app takes approximately 10-15 minutes to complete. The purpose of this study is to evaluate the efficacy of the Health-E You app among male youth ages 13-21 using a cluster-randomized stepped-wedge design. A participant will be considered to have completed the study if the participant has completed the baseline assessment, worked through the app, an immediate follow-up assessment, and a 2-month post-visit follow-up assessment. The end of the study is defined as completion of the 2-month follow-up assessment. Hypotheses include compared to usual care, app users will have greater improvements in male method use behaviors (i.e., condom use) as well as knowledge about pregnancy and sexually transmitted infection (STI) prevention methods, male method use self-efficacy, improved knowledge about SRH care, self-efficacy talking with a clinician about SRH, beliefs about SRH promotion, and SRH care receipt.

ELIGIBILITY:
Inclusion Criteria:

* Assigned male sex at birth
* Age 13 to 21 years old
* English and/or Spanish as preferred language to read, listen, and converse
* Self-reported engagement in vaginal and/or anal sex in the past 12 months
* Access to phone or internet for follow-up study activities

Exclusion Criteria:

* Aged 12 or younger or older than 21
* Primary language other than English or Spanish
* Not able to provide informed consent
* Unable to communicate due to cognitive, mental, language, or other difficulties
* Not sexually active, engaged in oral sex only, or more than 12 months have passed since last vaginal and/or anal sex.
* Previous participation in a Health-E You study activity or the app

Ages: 13 Years to 21 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2752 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Correct Condom Use Self-Efficacy Scale | Baseline, 24 hours after visit, 2-month follow-up
  Higher score indicates greater self-efficacy for correct use of male condoms. This measure is scaled with range from 1 (very difficult) to 5 (very easy); range 7-35.
Perceived efficacy in patient-physician interactions (PEPPI) | Baseline, 24 hours after visit, 2-month follow-up
  Higher score indicates greater efficacy in patient-physician interaction about sexual and reproductive health. This measure is scaled with range from 1 (not at all confident) to 5 (very confident); range 5-25.
Frequency condom use | Baseline, 2-month follow-up
  Measures frequency condom use with main & non-main partners in past year and last 2 months
Sexual and reproductive care receipt | Baseline, 24 hours after visit, 2-month follow-up
  Measures receipt of the recommended sexual and reproductive care package, based on national guidelines outlined by the Centers for Disease Control and Prevention (CDC) Office of Population Affairs (OPA) Quality Family Planning guidance & American Academy of Pediatrics' Bright Futures

CONTACTS AND LOCATIONS:
Overall Officials: Arik V Marcell, MD, MPH, Principal Investigator — Johns Hopkins Dept of Pediatrics / Division of Adolescent/Young Adult Medicine
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
The final version of collected data will be made available within thirty (30) months after the end of the data collection. Data will be preserved and made accessible along with the data codebook and other relevant documentation via the chosen repository. The investigators will make the data available through restricted/controlled access. Open Inter-university Consortium for Political and Social Research's (ICPSR's) Traditional Restricted Data or Physical Data Enclave will be used for some or all of the data, with restricted access solely to approved researchers.

REFERENCES:
- [Background] Akande M, Aturaliya R, Osio Smith S, Smith A, Arrington-Sanders R, Tebb K, Marcell AV. Integrating Young Male Voices to Enhance Sexual and Reproductive Healthcare Uptake of Innovative Pre-Clinic Technology. Journal of Adolescent Health. 2024;74(3 Suppl):S2.
- [Background] Tebb KP, Rodriguez F, Pollack LM, Adams S, Rico R, Renteria R, Trieu SL, Hwang L, Brindis CD, Ozer E, Puffer M. Improving contraceptive use among Latina adolescents: A cluster-randomized controlled trial evaluating an mHealth application, Health-E You/Salud iTu. Contraception. 2021 Sep;104(3):246-253. doi: 10.1016/j.contraception.2021.03.004. Epub 2021 Mar 17. PMID 33744300
- [Derived] Marcell AV, Smith AD, Osio Smith S, Akande M, Rohlff S, Arrington-Sanders R, Tebb K. A Previsit Mobile Health App (Health-E You/Salud iTu) for Male Adolescents to Promote Sexual and Reproductive Health Care Receipt: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2025 Oct 15;14:e77780. doi: 10.2196/77780. PMID 41092393